CLINICAL TRIAL: NCT00447902
Title: Safety and Antiviral Activity of TPV in Hepatitis C or Hepatitis B HIV Coinfected Patients - TDM Randomised Pilot Evaluation
Brief Title: Safety and Antiviral Activity of TPV in HCV and/or HBV HIV Coinfected Patients TDM Randomised Pilot Evaluation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 1182.99; EudraCT No.: 2005-005023-33
Record Dates: First submitted 2007-03-14; First posted 2007-03-15 (Estimated); Results first posted 2009-12-23 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections
Keywords: treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — tipranavir; Ritonavir

INTERVENTIONS:
Drug: tipranavir
Drug: ritonavir

SUMMARY:
The main purposes of this study are: demonstrate the safety and efficacy of TPV/r among HCV or hepatitis B virus (HBV) co-infected HIV+population, three-class (NRTI, NNRTI, and PI) experienced, with documented resistance to more than one PI. Determine pharmacokinetic data in this co-infected population and potential utility of using therapeutic drug monitoring (TDM) in improving efficacy outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected males or females at least 18 years of age.
2. Three-class (Nucleoside reverse transcriptase inhibitor (NRTI), Non nucleoside reverse transcriptase inhibitor (NNRTI), and Protease inhibitor (PI)) treatment-experienced (a minimum of 3-months duration for each class) with resistance to more than one PI (on the screening resistance testing). Patients that are NNRTI-naïve patients but who have genotypically documented NNRTI-resistance mutations on past or screening resistance testing would be eligible.
3. CD4+ T lymphocyte count ≥50 cells/µl and HIV-1 VL ≥1000 copies/mL at screening.
4. The ARV study treatment regimen must consist of new TPV/r in combination with an OBR of 2-4 agents of the following: N(t)RTIs (NRTI or NtRTI), enfuvirtide (ENF), and/or, where available, an Expanded Access Program (EAP) investigational agent (Section 3.3). In total, patients are to have an ARV study treatment regimen consisting of at least 3 agents (TPV/r and two OBRs).
5. Chronic hepatitis C Virus (HCV) infection demonstrated by HCV-ribonucleic acid (RNA) positivity or, Chronic hepatitis B (HB) infection demonstrated by anti HBc IgG Antibody and HB Surface Antigen positivity.
6. Acceptable screening laboratory values that indicate adequate baseline organ function.
7. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < Division of AIDS (DAIDS) Grade 3.
8. Acceptable medical history, as assessed by the investigator.
9. Any AIDS defining illness listed in the Appendix 10.3.1 should be accepted as long as is resolved, asymptomatic or stable on treatment for at least 12 weeks before screening (Visit 1); the AIDS defining events listed below are not acceptable History of Progressive Multifocal Leukoencephalopathy (PML), Visceral Kaposi's Sarcoma (KS), and/or any malignancy.
10. A reliable method of barrier contraception will be used by all female patients who are of reproductive potential, for at least three months prior to Visit 3, during the trial, and 30 days after completion or termination from the trial.
11. Karnofsky performance score ≥70.

Exclusion Criteria:

1. Prior tipranavir use.
2. Known hypersensitivity to any of the ingredients to the tipranavir or ritonavir formulations.
3. ARV medication naive.
4. Genotypic resistance to Tipranavir (TPV) (defined as a TPV mutation score of more than 7).
5. Patients on recent drug holiday, defined as off ARV medications for at least 7 consecutive days within the month prior to screening.
6. Decompensated liver disease, including presence or history of ascites, variceal bleeding, or hepatic encephalopathy or having ever been diagnosed as having hepatic insufficiency of Child Pugh class B or C.
7. Female patients of childbearing potential who:

   * have a positive serum pregnancy test at screening,
   * are breast feeding,
   * are planning to become pregnant,
   * are not willing to use a barrier method of contraception, or
   * are only willing to use an estrogen-containing medication, e.g., ethinyl estradiol, as a method of contraception.
8. Use of investigational medications within 30 days before study entry or during the trial except for those investigational ARV drugs permitted during the trial as stated in inclusion criteria 6.
9. Use of concomitant drugs that may significantly reduce plasma levels of the study medications.
10. Use of immunomodulatory drugs or antineoplastic agents within 30 days before study entry or during the trial.
11. Inability to adhere to the requirements of the protocol, including active substance abuse, as defined by the investigator.
12. Anticipated need for an interferon-based regimen in the 48 weeks following the study entry.
13. Any other or additional plausible cause for chronic liver disease, including the presence of other viruses known or suspected to cause hepatitis.
14. Any active infection or neoplasm currently being treated.
15. Patients with history of hemorrhagic stroke or intracranial aneurysm.
16. Patients with history of ischemic stroke, neurosurgery, skull trauma and/or intracranial pathology (arteriovenous malformation, brain tumors and cerebral venous thrombosis) within 4 weeks prior to screening (Visit 1) as assessed by investigator.
17. Patients with current history of alcohol abuse defined as alcohol consumption that would interfere with patient's compliance or result in biological abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (30):
- United States (5):
  - 1182.99.32 Boehringer Ingelheim Investigational Site, Beverly Hills, California
  - 1182.99.31 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1182.99.12 Boehringer Ingelheim Investigational Site, Providence, Rhode Island
  - 1182.99.1 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1182.99.4 Boehringer Ingelheim Investigational Site, Houston, Texas
- 1182.99.54001, Capital Federal, Argentina
- Brazil (4):
  - 1182.99.55002 Hospital DIA, Sacomã - São Paulo
  - 1182.99.55004 Unidade de Referência em doenças Infecciosas Preveníveis, Santo André
  - 1182.99.55001 Universidade Federal de Sao Paulo, São Paulo
  - 1182.99.55003 Centro de Referência e Treinamento - DST/AIDS, Vila Mariana - Sao Paulo
- France (12):
  - 1182.99.3301A Boehringer Ingelheim Investigational Site, Garches
  - 1182.99.3306G Boehringer Ingelheim Investigational Site, Nantes
  - 1182.99.3306K Boehringer Ingelheim Investigational Site, Nantes
  - 1182.99.3310C Boehringer Ingelheim Investigational Site, Nice
  - 1182.99.3310D Boehringer Ingelheim Investigational Site, Nice
  - 1182.99.3310E Boehringer Ingelheim Investigational Site, Nice
  - 1182.99.3310F Boehringer Ingelheim Investigational Site, Nice
  - 1182.99.3310G Boehringer Ingelheim Investigational Site, Nice
  - 1182.99.3310H Boehringer Ingelheim Investigational Site, Nice
  - 1182.99.3304A Boehringer Ingelheim Investigational Site, Paris
  - 1182.99.3304C Boehringer Ingelheim Investigational Site, Paris
  - 1182.99.3302A Boehringer Ingelheim Investigational Site, Perpignan
- 1182.99.4909 Boehringer Ingelheim Investigational Site, Düsseldorf, Germany
- Italy (5):
  - 1182.99.3912 Boehringer Ingelheim Investigational Site, Ancona
  - 1182.99.3901 Boehringer Ingelheim Investigational Site, Milan
  - 1182.99.3911 Boehringer Ingelheim Investigational Site, Milan
  - 1182.99.3916 Boehringer Ingelheim Investigational Site, Milan
  - 1182.99.3906 Boehringer Ingelheim Investigational Site, Pavia
- Spain (2):
  - 1182.99.3402, Barcelona
  - 1182.99.3407, Madrid

RESULTS

PARTICIPANT FLOW:
Recruitment Details: With FDA and EMEA agreement, the trial was prematurely discontinued before reaching the target number of patients to be entered due to poor recruitment. For this reason analyzing and reporting data as planned for primary and secondary endpoints have not been performed. No objectives were reached and no conclusion can be drawn from this study.
Pre-assignment Details: One patient has been randomised by mistake in Brasil and so he was not treated
Groups:
- Standard of Care: Tipranavir (TPV) 500mg and Ritonavir (RTV) 200mg BID capsules
- Therapeutic Drug Monitoring: Tipranavir (TPV) 500mg and Ritonavir (RTV) 200mg BID capsules as initial dose, increased to TPV/r 750mg/200mg BID capsules, or decreased to TPV/r 500mg/100mg BID capsules or TPV/r 250mg/200mg BID capsules
Period: Overall Study
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Started | 5 | 6
Completed | 1 | 0
Not Completed | 4 | 6
Not completed — Adverse Event | 0 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — included patients who discontinued | 1 | 1
Not completed — Lack of Efficacy | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Therapeutic Drug Monitoring | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.00 (2.90) | 45.20 (5.40) | 45.50 (4.40)
Sex: Female, Male [Count of Participants; unit: Participants] — Included patients who discontinued due to early termination
  Participants
    Female | 1 | 1 | 2
    Male | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response at Week 48
Description: Treatment response is a confirmed virologic response, defined as a viral load less than 50 copies/mL at two consecutive measurements at least 5 days apart, without death, permanent discontinuation, or introduction of a new antiretroviral
Time Frame: 48 weeks
Population: The trial has been stopped due to a poor enrollment
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Virologic Response Defined as Viral Load <50 Copies/mL at Each Visit
Description: Virologic response defined as viral load less than 50 copies/mL
Time Frame: After 4 weeks of treatment until the end of the trial
Population: The trial has been stopped due to a poor enrollment
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Occurrence of Viral Load Less Than 400 Copies/mL at Weeks 24 and 48
Description: Patients with a viral load of less than 400 copies/mL at Weeks 24 and 48 as measured from a plasma sample.
Time Frame: 24 and 48 weeks
Population: The trial has been stopped due to a poor enrollment
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Occurrence of Viral Load Less Than 400 Copies/mL at Each Visit
Description: Patients with a viral load of less than 400 copies/mL at each visit as measured from a plasma sample.
Time Frame: After 4 weeks of treatment until the end of the trial
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Occurrence of ≥1 log10 Drop in Viral Load From Baseline at All Visits, Including Visits at Weeks 24 and 48
Description: Occurrence of greater than or equal to 1 log10 drop in viral load from baseline at all visits, including visits at Weeks 24 and 48
Time Frame: Baseline, 24 and 48 weeks
Population: The trial has been stopped due to a poor enrollment
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Viral Load From Baseline at Each Visit
Description: Change in viral load (measured from a plasma sample) from baseline at each visitPatients with a viral load of less than 400 copies/mL at each visit as .
Time Frame: After 4 weeks of treatment until the end of the trial
Population: The trial has been stopped due to a poor enrollment
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Time to Treatment Failure
Description: For patients who never achieve a confirmed virologic response, time to treatment failure is defined as 0. For patients who achieve a confirmed virologic response, time to treatment failure is the earliest time of either: death, permanent discontinuation of the study drug or loss to follow-up, introduction of a new anti-retroviral drug to the regimen if it is not solely related to either toxicity or intolerance clearly attributable to a background drug, but not the study drug, or first occurrence of a VL >50 copies/mL at two consecutive measurements after having achieved a VL <50 copies/mL.
Time Frame: After Day 1 of treatment until the end of the trial
Population: The trial has been stopped due to a poor enrollment
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Time to New AIDS or AIDS Related Progression Event or Death
Description: Time to new AIDS or AIDS related progression event or death as defined by AIDS defining and/or AIDS-related illnesses.
Time Frame: After Day 1 of treatment until the end of the trial
Population: The trial has been stopped due to a poor enrollment
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in CD4+ and CD8+ Cell Counts From Baseline to Week 48
Description: Change from baseline to Week 48 for CD4+ and CD8+ cell counts. Samples were obtained for CD4+ and CD8+ as measurements of viral suppression during antiretroviral therapy.
Time Frame: after 2 weeks of treatment till Week 48
Population: The trial has been stopped due to a poor enrollment
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in Ratio of CD38+/CD8+ From Baseline to Week 48
Description: Change from baseline to Week 48 for the ratio of CD38+ to CD8+ cell counts. Samples were obtained for CD38+ and CD8+ as measurements of viral suppression during antiretroviral therapy.
Time Frame: after 2 weeks of treatment till Week 48
Population: The trial has been stopped due to a poor enrollment
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in Ratio of CD3+ CD8+ CD38+ HLA DR From Baseline to Week 48.
Description: Change from baseline to Week 48 for the ratio of CD3+ CD8+ CD38+ HLA DR . Samples were obtained for CD3+ CD8+ CD38+ HLA DR as measurements of viral suppression during antiretroviral therapy.
Time Frame: after 2 weeks of treatment till Week 48
Population: The trial has been stopped due to a poor enrollment
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Tipranavir (TPV) and Ritonavir (RTV) Trough Concentrations at Week 2, Week 4, Week 8, Week 12, Week 24, Week 36 and Week 48
Description: Tipranavir (TPV) and Ritonavir (RTV) trough concentrations from plasma samples at Week 2, Week 4, Week 8, Week 12, Week 24, Week 36 and Week 48
Time Frame: after 2 weeks of treatment till Week 48
Population: The trial has been stopped due to a poor enrollment
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Patients Adherence With Study Medication Based on Pill Count
Description: number of pills actually taken divided by the planned number of pills the patient should take
Time Frame: After 4 weeks of treatment until the end of the trial
Population: The trial has been stopped due to a poor enrollment
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Occurrence of Tipranavir (TPV) Inhibitory Quotient (IQ) >60 at Each Visit Where TPV Concentration is Measured
Description: A high inhibitory quotient (IQ), the ratio of trough plasma drug concentration to the protein-adjusted viral IC50, is a useful indicator of the potential efficacy margin of antiretroviral drugs. The IQ for TPV is calculated by the formula IQ = TPV Ctrough / (3.75 x Z x fold change of the patients virus), where Z = wild type control IC50 IIIB.
Time Frame: After 2 weeks of treatment until the end of trial
Population: The trial has been stopped due to a poor enrollment
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Occurrence of Tipranavir (TPV) Trough Concentration >120 μM
Description: Patients with TPV trough above 120 μM are at high risk of developing a Grade 3 or 4 ALT or AST elevations. The risk of Grade 3 or greater transaminase elevations appeared to be uniform at TPV trough concentration below 120 μM. Hence, for this study the TPV trough should be maintained below 120 μM.
Time Frame: After 2 weeks of treatment until the end of trial
Population: The trial has been stopped due to a poor enrollment
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Post-dose Tipranavir (TPV) and Ritonavir (RTV) Concentrations at Week 4
Description: Post-dose Tipranavir (TPV) and Ritonavir (RTV) plasma concentrations at Week 4
Time Frame: Week 4
Population: The trial has been stopped due to a poor enrollment
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Frequency of Patients (%) With Possible Clinically Significant Abnormalities of Laboratory Measurements
Description: Frequency of patients (%) with possible clinically significant abnormalities of laboratory measurements (haematology, differentials (automatic and absolute), coagulation, electrolytes, enzymes, substrates, urinalysis, serology and T-cells)
Time Frame: Baseline through 48 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Number analyzed (Participants) | 4 | 6
percentage of participants
  Hematocrit - decrease | 25.0 | 16.7
  Red Blood Cell count - decrease | 25.0 | 0
  Prothrombin time - increase | 0 | 20.0
  AST/GOT, SGOT - increase | 50.0 | 33.3
  ALT/GPT, SGPT - increase | 25.0 | 33.3
  Lipase - increase | 0 | 16.7
  Bilirubin, total - increase | 0 | 16.7
  Bilirubin, direct - increase | 0 | 16.7
  Triglyceride - increase | 0 | 25.0

18. Primary Outcome: The Primary Safety Endpoint Was the Occurrence of Dose-limiting Hepatotoxicity During the Study.
Description: Dose-limiting hepatotoxicity was defined as Grade 4 ALT or AST elevation confirmed in 48h or any evocative symptoms or signs of hepatitis, if it not clearly attributable to another cause. Patients who experienced dose-limiting hepatotoxicity stopped TPV/r and were considered treatment failures for the analysis.
Time Frame: From the start of the study through 48 weeks.
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening through the duration of the trial (Week 48 planned).
Arm/Group | Standard of Care | Therapeutic Drug Monitoring
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/6
Other Adverse Events (participants affected / at risk) | 3/4 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=4) | Therapeutic Drug Monitoring (N=6)
pyrexia (General disorders) | 1 | 0
cardio respiratory arrest (Cardiac disorders) | 0 | 1
abdominal pain (Gastrointestinal disorders) | 0 | 1
abdominal pain upper (Gastrointestinal disorders) | 0 | 1
diarrhoea (Gastrointestinal disorders) | 0 | 1
faeces discoloured (Gastrointestinal disorders) | 0 | 1
vomiting (Gastrointestinal disorders) | 0 | 1
cholelithiasis (Hepatobiliary disorders) | 0 | 1
aspartate aminotransferase increased (Investigations) | 0 | 1
alanine aminotransferase increased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=4) | Therapeutic Drug Monitoring (N=6)
oral candidiasis (Infections and infestations) | 1 | 0
sinusitis (Infections and infestations) | 1 | 0
hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
dizziness (Nervous system disorders) | 0 | 1
headache (Nervous system disorders) | 0 | 1
paraesthesia (Nervous system disorders) | 0 | 1
vertigo (Ear and labyrinth disorders) | 0 | 1
palpitations (Cardiac disorders) | 0 | 1
abdominal pain (Gastrointestinal disorders) | 1 | 0
dysphagia (Gastrointestinal disorders) | 1 | 0
erythema (Skin and subcutaneous tissue disorders) | 0 | 1
back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
adverse drug reaction (General disorders) | 2 | 0
pyrexia (General disorders) | 1 | 0
fatigue (General disorders) | 1 | 0
injection site nodule (General disorders) | 1 | 0
nodule (General disorders) | 1 | 0
alanine aminotransferase increased (Investigations) | 0 | 1
blood albumin decreased (Investigations) | 1 | 0
haemoglobin decrease (Investigations) | 1 | 0
Skin nodules (Skin and subcutaneous tissue disorders) | 1 | 0
aspartate aminotransferase increased (Investigations) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to an early termination of the trial no analysis has been performed for primary and secondary endpoints

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.